CLINICAL TRIAL: NCT07054697
Title: A Single-blind Randomized Placebo Controlled Pilot Study With Individualized Homeopathic Treatment in the Children With Autism Spectrum Disorder
Brief Title: Pilot-RCT With Individualized Homeopathic Treatment in the Children With Autism Spectrum Disorder
Acronym: Pilot-RCT ASD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aditi Chadha (Other)
Responsible Party: Sponsor-Investigator, Aditi Chadha, DOCTOR, Tatva Homoeopathic Clinic and Research Centre
Organization: Tatva Homoeopathic Clinic and Research Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20172024
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: Homoeopathy; Autism Spectrum Disorder; Randomized Controlled Trial
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Homeopathy; Smallpox Vaccine; Causticum; Tuberculin; Datura stramonium lectin; Calcium Carbonate; Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HOMOEOPATHIC GROUP (Experimental)
  Interventions: Drug: Homoeopathic medicines; Behavioral: THERAPY
- CONTROL GROUP (Placebo Comparator): SACCHARUM LACTIS
  Interventions: Drug: Placebo; Behavioral: THERAPY

INTERVENTIONS:
Drug: Homoeopathic medicines
  Other Names: THUJA OFFICINALIS; VACCININUM; CAUSTICUM; ARGENTUM NITRICUM; TUBERCULINUM; STRAMONIUM; STAPHYSAGRIA; ARUM TRIPHYLLUM; BACILLINUM; CINA; CARCINOCIN; CUPRUM METALLICUM; AMBER GRISEA; CALCAREA CARBONICA; CROCUS SATIVUS; HEPAR SULPHUR; HYOSCYMUS; KALI BROMATUM; LAC VACCININUM; MEDORRHINUM; NATRUM PHOSPHORICUM
  Arms: HOMOEOPATHIC GROUP
Drug: Placebo
  Other Names: SACCHARUM LACTIS
  Arms: CONTROL GROUP
Behavioral: THERAPY — SPEECH THERAPY / OCCUPATIONAL THERAPY

SUMMARY:
This study looked at whether homeopathic treatment could help children with Autism Spectrum Disorder (ASD) when used alongside regular therapies like speech and occupational therapy. Over seven years, children between the ages of 2 and 12 were divided into two groups (through computer generated list). One group received individualized homeopathic medicines, and the other received a look-alike placebo (with no active ingredients). Meanwhile, both the groups continued with their regular therapies.

Researchers used various tools and parent questionnaires to track the children's progress in areas like communication, behavior, social skills, daily functioning, toilet training and sensory skills. They found that the children who received homeopathic treatment showed more improvement in these areas compared to those who just received only speech / occupational therapies.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of Autism Spectrum Disorder (ABC score ≥ 67)
* Age range of 2 to 12 years

Exclusion Criteria:

* Children with other significant comorbid psychiatric conditions that could confound the results. [eg. a brain injury; fragile X syndrome or other syndromes resulting from known genetic defects or inherited metabolic diseases; other diagnosed conditions involving impairments in social and communication abilities, such as intellectual disability without ASD, schizophrenia, language disorders and social communication disorder]
* Children with irregular follow ups.
* Children with poor medical compliance.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Childhood Autism Rating Scale (CARS) | BASELINE, YEARLY (0-7 YEARS)
  To measure various behavioral dimensions and adaptive functioning
Autism Treatment Evaluation Checklist (ATEC) | BASELINE, YEARLY (0 - 7 YEARS)
  To assess the efficacy of the treatment among both the arms.

SECONDARY OUTCOMES:
Social Responsiveness Scale (SRS) | BASELINE, YEARLY (0 - 7 YEARS)
  To measure social skills, communication abilities.
Neurodevelopmental Parent Report for Outcome Monitoring (ND PROM) | BASELINE, YEARLY (0 - 7 YEARS)
  To gather subjective reports on their children's behavior, social interactions, and overall well-being from the parents.

CONTACTS AND LOCATIONS:
Locations (1):
- Holistic Homoeopathic Clinic and Research Center, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided
TO MAINTAIN CONFIDENTIALITY